CLINICAL TRIAL: NCT03833388
Title: A Multi-Center, Randomized, Double Masked, Placebo Controlled Clinical Study to Assess the Efficacy and Safety of TOP1630 0.1% Ophthalmic Solution Compared to Placebo in Subjects With Moderate to Severe Dry Eye Syndrome
Brief Title: Study of TOP1630 for Dry Eye Syndrome
Acronym: THEIA-1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Topivert Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOP1630-TV-05
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TOP1630 Ophthalmic Solution (Experimental)
  Interventions: Drug: TOP1630 0.1% Ophthalmic Solution TID OU
- Placebo to TOP1630 Ophthalmic Solution (Placebo Comparator)
  Interventions: Drug: Placebo to TOP1630 0.1% Ophthalmic Solution TID OU

INTERVENTIONS:
Drug: TOP1630 0.1% Ophthalmic Solution TID OU — Bilateral ocular drug administration
  Arms: TOP1630 Ophthalmic Solution
Drug: Placebo to TOP1630 0.1% Ophthalmic Solution TID OU — Bilateral ocular drug administration
  Arms: Placebo to TOP1630 Ophthalmic Solution

SUMMARY:
In subjects with Dry Eye Syndrome (DES):

The primary objective of this study is to confirm the efficacy of TOP1630 0.1% Ophthalmic Solution TID OU compared to placebo treatment at Day 29 on pre-specified sign and symptom endpoints in subjects with moderate to severe DES.

DETAILED DESCRIPTION:
This study is designed to assess the efficacy and safety of TOP1630 ophthalmic solution in subjects with Dry Eye Syndrome (DES).

Eligible subjects will be randomized double masked to either TOP1630 or placebo for a duration of 28 days' treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a reported history of dry eye;
* Have a history of use of eye drops for dry eye symptoms;

Symptoms of dry eye syndrome including:

* Ocular discomfort
* Conjunctival redness
* Tear film break up time
* Schirmer test score

Signs of dry eye syndrome including:

* Conjunctival staining score

Exclusion Criteria:

* Have any clinically significant slit lamp findings at entry visit ;
* Be diagnosed with an ongoing ocular infection;
* Have any significant ocular lesion that could interfere with assessment of safety or efficacy or prevent study conduct in the opinion of the PI;
* Have any planned ocular and/or lid surgeries over the study period;
* Have an uncontrolled systemic disease;
* Be a woman who is pregnant, nursing or planning a pregnancy;
* Be a woman of childbearing potential who is not using an acceptable means of birth control;
* Have a known allergy and/or sensitivity to the test article or its components;
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Ocular grittiness 6-point (0-5) scale | Day 29
  Ocular grittiness severity assessment
Ocular surface (all-regions) lissamine green staining score 5-point (0-4) scale each region | Day 29
  Dry Eye Syndrome ocular staining assessment. Total region score: inferior, superior, central, temporal, and nasal.

SECONDARY OUTCOMES:
Ocular discomfort 5-point (0-4) scale | Day 29
  Ocular discomfort severity assessment
Ocular dryness 6-point (0-5) scale | Day 29
  Ocular dryness severity assessment
Conjunctival lissamine green staining score 5-point (0-4) scale each region | Day 29
  Dry Eye Syndrome ocular staining assessment. Conjunctival sum score: temporal and nasal.
Corneal lissamine green staining score 5-point (0-4) scale each region | Day 29
  Dry Eye Syndrome ocular staining assessment. Corneal sum score: inferior, superior and central.
Worst ocular symptom 6-point (0-5) scale | Day 29
  Most severe baseline symptom from reported daily symptoms

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Central Maine Eye Care, Lewiston, Maine
  - Andover Eye Associates, Andover, Massachusetts
  - Suite 305, 775 Paramount Drive, Raynham, Massachusetts
  - Total Eye Care, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided